CLINICAL TRIAL: NCT04231539
Title: Pharmacokinetics, Subjective Effects, and Abuse Liability of Nicotine Salt-Based Vaping Products With Tobacco or Unflavored E-liquids[SALTVAPE Study]
Brief Title: Pharmacokinetics, Subjective Effects, and Abuse Liability of Nicotine Salt-Based Vaping Products With Tobacco or Unflavored E-liquids, SALTVAPE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: I 475819; NCI-2019-07370 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 475819 (Other: Roswell Park Cancer Institute); U54CA228110 (NIH)
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: The participant and researcher will be blinded to solution flavor and nicotine concentrates.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (14):
- Product Sequence D (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Device: Vaporizer Device; Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product Sequence A then B then C (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C)
- Product sequence B then C then A then D (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence D then B then A then C (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence C then D then B then A (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence A then C (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Free-Low Nicotine Tobacco Flavored (Product C)
- Product sequence D then C then B then A (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence A then D then B then C (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence D then A then C then B (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence C then D then A then B (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence A then C then D then B (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product Sequence A then B then D then C (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence B then A then D thn C (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)
- Product sequence B then D then C then A (Experimental): After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt based nicotine e-liquid solution of tobacco flavor assigned in a random order.
  Interventions: Drug: Nicotine; Device: Vaporizer Device; Drug: Salt-HIgh Nicotine Unflavored (Product B); Drug: Free-Low Nicotine Tobacco Flavored (Product C); Drug: Salt-High Nicotine Tobacco Flavored (Product D)

INTERVENTIONS:
Drug: Nicotine — Vape Free-Low nicotine unflavored
  Other Names: Free-Low Nicotine Unflavored (Product A); NIC
  Arms: Product Sequence A then B then C; Product Sequence A then B then D then C; Product sequence A then C; Product sequence A then C then D then B; Product sequence A then D then B then C; Product sequence B then A then D thn C; Product sequence B then C then A then D; Product sequence B then D then C then A; Product sequence C then D then A then B; Product sequence C then D then B then A; Product sequence D then A then C then B; Product sequence D then B then A then C; Product sequence D then C then B then A
Device: Vaporizer Device — Take puffs from vaporizer filled with different flavors
  Other Names: Vaporizer
Drug: Salt-HIgh Nicotine Unflavored (Product B) — Vape Salt-High nicotine unflavored
  Arms: Product Sequence A then B then C; Product Sequence A then B then D then C; Product sequence A then C then D then B; Product sequence A then D then B then C; Product sequence B then A then D thn C; Product sequence B then C then A then D; Product sequence B then D then C then A; Product sequence C then D then A then B; Product sequence C then D then B then A; Product sequence D then A then C then B; Product sequence D then B then A then C; Product sequence D then C then B then A
Drug: Free-Low Nicotine Tobacco Flavored (Product C) — Vape Free-Low Nicotine Tobacco
  Arms: Product Sequence A then B then C; Product Sequence A then B then D then C; Product sequence A then C; Product sequence A then C then D then B; Product sequence A then D then B then C; Product sequence B then A then D thn C; Product sequence B then C then A then D; Product sequence B then D then C then A; Product sequence C then D then A then B; Product sequence C then D then B then A; Product sequence D then A then C then B; Product sequence D then B then A then C; Product sequence D then C then B then A
Drug: Salt-High Nicotine Tobacco Flavored (Product D) — Vape Salt-High Tobacco
  Arms: Product Sequence A then B then D then C; Product Sequence D; Product sequence A then C then D then B; Product sequence A then D then B then C; Product sequence B then A then D thn C; Product sequence B then C then A then D; Product sequence B then D then C then A; Product sequence C then D then A then B; Product sequence C then D then B then A; Product sequence D then A then C then B; Product sequence D then B then A then C; Product sequence D then C then B then A

SUMMARY:
This trial studies activity of time (pharmacokinetics), subjective effects, and abuse liability of nicotine salt-based vaping products with tobacco or e-liquids. This study aims to determine and compare the levels of nicotine delivered to the bloodstream from nicotine salt and free-base nicotine e-liquid solutions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of nicotine salt (nicotine benzoate) and free-base nicotine in different flavored e-liquid solutions on puffing behaviors and systemic exposure to nicotine from electronic nicotine delivery systems (ENDS) by:

Ia. Assessing short-term effects on nicotine cravings, withdrawal, and satisfaction from single use of ENDS refilled with flavored nicotine salt or flavored free-base nicotine solutions with two different flavors (tobacco or unflavored) in current daily ENDS users following an overnight fast.

Ib. Comparing users' perceptions and preferences towards inhaling vapors containing nicotine salt (nicotine benzoate) or freebase nicotine with two different flavors (tobacco and unflavored) versus their regular brand.

II. This project provides important information on whether the pharmacokinetics of nicotine delivery differ between salt and free-base forms of e-liquid of equivalent nominal concentration using the same device, and whether the previously observed effects of flavors on subjective effects differ between salt and free-base forms.

III. Determine whether maximum concentration of nicotine in plasma (Cmax) or time to maximum concentration (Tmax) differ between free-base and salt-based versions of the same liquid, controlling for flavoring and nominal nicotine concentration [main effect of salt].

IV. Determine whether the effect of flavoring on subjective effects (e.g., harshness, liking) differs between matched free-base and salt-based e-liquids [flavor X salt interaction].

EXPLORATORY OBJECTIVE:

I. Examine effects of salt and flavoring on abuse liability using the Experimental Tobacco Marketplace (ETM).

OUTLINE:

After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours, 5-7 days apart. During each session, participants take 20 puffs over 10 minutes (one puff every 30 seconds) of vaporizer filled with freebased nicotine electronic (e)-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored, or salt-based nicotine e-liquid solution of tobacco flavor assigned in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to abstain from using ENDS product for 8-10 hours (overnight abstinence) prior to study visits
* Current daily ENDS user as determined by

  * Has used ENDS product every day for the past 6 months (by history)
  * Has used ENDS product or e-liquid containing nicotine (by history)
* Participant or legal representative must understand the investigational nature of this study and sign and Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Smoked cigarettes in the past 7 days
* Currently smokes >= 5 cigarettes per month
* Unstable medical conditions (such as unstable heart disease, uncontrolled hypertension, thyroid disease, diabetes, renal or liver impairment, or glaucoma) or psychiatric condition (such as current major depression, history of schizophrenia or bipolar disorder) or current regular use of psychiatric medications (such as major tranquilizers and antidepressants)
* History of serious side effects from nicotine or from any nicotine replacement therapies
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing females
* Concurrent participation in another clinical trial
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Quisenberry, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Product Sequence D: After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with one of the following: freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt-based nicotine e-liquid solution of tobacco flavor assigned in random order.
  Vaporizer Device: Take puffs from vaporizer filled with different flavors
  Salt-High Nicotine Tobacco Flavored (Product D): Vape Salt-High Tobacco
- Product Sequence A then B then C: After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with one of the following: freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt-based nicotine e-liquid solution of tobacco flavor assigned in random order.
  Nicotine: Vape Free-Low nicotine unflavored
  Vaporizer Device: Take puffs from vaporizer filled with different flavors
  Salt-HIgh Nicotine Unflavored (Product B): Vape Salt-High nicotine unflavored
  Free-Low Nicotine Tobacco Flavored (Product C): Vape Free-Low Nicotine Tobacco
- Product sequence B then C then A then D; Product sequence D then B then A then C; Product sequence C then D then B then A; Product sequence D then C then B then A; Product sequence A then D then B then C; Product sequence D then A then C then B; Product sequence C then D then A then B; Product sequence A then C then D then B; Product Sequence A then B then D then C; Product sequence B then A then D thn C; Product sequence B then D then C then A: After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with one of the following: freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt-based nicotine e-liquid solution of tobacco flavor assigned in random order.
  Nicotine: Vape Free-Low nicotine unflavored
  Vaporizer Device: Take puffs from vaporizer filled with different flavors
  Salt-HIgh Nicotine Unflavored (Product B): Vape Salt-High nicotine unflavored
  Free-Low Nicotine Tobacco Flavored (Product C): Vape Free-Low Nicotine Tobacco
  Salt-High Nicotine Tobacco Flavored (Product D): Vape Salt-High Tobacco
- Product sequence A then C: After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with one of the following: freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt-based nicotine e-liquid solution of tobacco flavor assigned in random order.
  Nicotine: Vape Free-Low nicotine unflavored
  Vaporizer Device: Take puffs from vaporizer filled with different flavors
  Free-Low Nicotine Tobacco Flavored (Product C): Vape Free-Low Nicotine Tobacco
Period: Overall Study
Arm/Group | Product Sequence D | Product Sequence A then B then C | Product sequence B then C then A then D | Product sequence D then B then A then C | Product sequence C then D then B then A | Product sequence A then C | Product sequence D then C then B then A | Product sequence A then D then B then C | Product sequence D then A then C then B | Product sequence C then D then A then B | Product sequence A then C then D then B | Product Sequence A then B then D then C | Product sequence B then A then D thn C | Product sequence B then D then C then A
Started | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Product Sequence B Then C Then A Then D: After 8-10 hours after nicotine abstinence, participants attend 4 vaping sessions over 2-2.5 hours , 5-7 days apart. They are randomized to take 20 puffs over 10 minutes (1 puff every 30 seconds) of vaporized filled with one of the following: freebased nicotine e-liquid solution of unflavored, free-based nicotine e-liquid solution of tobacco flavor, salt-based nicotine e-liquid solution of unflavored or salt-based nicotine e-liquid solution of tobacco flavor assigned in random order.
  Vaporizer Device: Take puffs from vaporizer filled with different flavors
  Salt-HIgh Nicotine Unflavored (Product B): Vape Salt-High nicotine unflavored
  Free-Low Nicotine Tobacco Flavored (Product C): Vape Free-Low Nicotine Tobacco
  Salt-High Nicotine Tobacco Flavored (Product D): Vape Salt-High Tobacco
- Total: Total of all reporting groups
Arm/Group | Product Sequence D | Product Sequence A Then B Then C | Product Sequence B Then C Then A Then D | Product Sequence D Then B Then A Then C | Product Sequence C Then D Then B Then A | Product Sequence A Then C | Product Sequence D Then C Then B Then A | Product Sequence A Then D Then B Then C | Product Sequence D Then A Then C Then B | Product Sequence C Then D Then A Then B | Product Sequence A Then C Then D Then B | Product Sequence A Then B Then D Then C | Product Sequence B Then A Then D Thn C | Product Sequence B Then D Then C Then A | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (2.8) | 24 (na) — 1 observation | 55 (na) — 1 observation | 37 (na) — 1 observation | 21 (na) — 1 observation | 21 (na) — 1 observation | 24 (na) — 1 observation | 23 (na) — 1 observation | 29 (na) — 1 observation | 26 (na) — 1 observation | 22 (na) — 1 observation | 32 (na) — 1 observation | 33 (na) — 1 observation | 32 (na) — 1 observation | 28.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5
  Male | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration of Nicotine in Plasma (Cmax)
Description: The maximum nicotine concentration in blood plasma
Time Frame: Samples were taken at minutes 0, then they started puffing and samples were taken 2, 4, 5, 6, 8, 10 minutes during puffing. Then, samples were taken at times 13, 15, 20, 30, and 120 minutes post puffing. The last dose occurred at week 4.
Population: All treated and eligible patients
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- A: Unflavored Free-based Nicotine Form: Participants will sample a standardized e-cigarette with a formulation that contains free-based nicotine that is unflavored.
- B: Unflavored Salt-based Nicotine Form: Participants will sample a standardized e-cigarette with a formulation that contains salt-based nicotine that is unflavored.
- C: Tobacco Flavor Free-based Nicotine Form: Participants will sample a standardized e-cigarette with a formulation that contains free-based nicotine that is tobacco flavored.
- D: Tobacco Flavor Salt-based Nicotine Form: Participants will sample a standardized e-cigarette with a formulation that contains salt-based nicotine that is tobacco flavored.
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
ng/mL | 5.7 (0.8) | 11.8 (3.3) | 6.7 (1.3) | 8.1 (1.7)

2. Primary Outcome: Area Under the Concentration-time Curve (AUC)
Description: Area under the plasma nicotine concentration over time curve
Time Frame: as for outcome 1
Population: All treated and eligible patients
Measure: Mean (Standard Error); unit: ng*min/mL
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
ng*min/mL | 128.8 (40.8) | 295.6 (126.7) | 177.3 (51.7) | 199.7 (71.7)

3. Primary Outcome: Time to Maximum Concentration
Description: Time to maximum nicotine concentration in the blood plasma
Time Frame: as for outcome 1
Population: All treated and eligible patients
Measure: Mean (Standard Error); unit: minutes
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
minutes | 11.5 (1.6) | 9.8 (1.5) | 11.7 (1.5) | 8.6 (1.3)

4. Secondary Outcome: Perceived Harshness of Experimental Product Sampled
Description: Subjective Measure of Perceived Harshness (Likert, 1-5: 1 = best outcome, 5 = worst outcome).
Time Frame: 1 minute post puffing for 4 weeks
Population: All treated and eligible patients
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | 4.85 (0.1) | 2.92 (0.4) | 4.62 (0.1) | 3.08 (0.4)

5. Secondary Outcome: Perceived Satisfaction of Experimental Product Sampled
Description: Nicotine Solution Rating Scale that orders each of the four products from 1 to 4, with 1 being least satisfying and 4 being most satisfying. Mean rank is provided with a possible score of 1 through 4.
Time Frame: 120 minutes after session start on last session (session 4)
Population: All treated and eligible patients
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | 3.08 (0.3) | 3.75 (0.4) | 3.77 (0.4) | 4.23 (0.3)

6. Secondary Outcome: Perceived Liking of Experimental Product Sampled
Description: Drug Effects Questionnaire Item #1 - perceived liking of the experimental product assessed by the question, "Do you like any of the effects you are feeling right now?" on a Likert scale from 0 (not at all) to 100 (extremely), with lower scores representing less liking of the experimental product. Mean is provided with possible scores between 0 and 100.
Time Frame: 1 minute post puffing for 4 weeks
Population: All treated and eligible patients
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | 45.9 (5.2) | 55.2 (4.0) | 46.5 (6.0) | 52.5 (5.4)

7. Secondary Outcome: Minnesota Nicotine Withdrawal Scale Change (Change From Pre- to Post-)
Description: Minnesota Nicotine Withdrawal Scale Change
  Minnesota Nicotine Withdrawal scale measures 8 facets of withdrawal and results in a total score. We use change from 5 minutes Pre-puffing to 3 minutes post puffing session. Individual questions are scored 0 (none/better) to 4 (severe/worse). And then the scores are totaled. Positive change score = more withdrawal symptoms. Change score can range from -32 to 36).
  Positive change score = worse withdrawal symptoms
  Individual questions are scored 0 (none/better) to 4 (severe/worse). And then the scores are totaled.
Time Frame: 5 minutes pre puffing and 3 minutes post puffing for 4 weeks
Population: All treated and eligible patients
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | 0.5 (0.7) | 0.7 (0.7) | 1.5 (0.5) | -0.5 (0.7)

8. Other Pre Specified Outcome: Intensity of Demand or Estimated Milligrams E-cigarettes Purchased at Free Cost for Each Device Sampled
Description: Demand intensity is a behavioral economic estimated measure of consumption at zero cost in a experimental marketplace focused on purchasing of tobacco and nicotine products over increasing price of one product while others stay the same price. Participants were asked to purchase tobacco products (12 options) for one week's use. At each of the four sessions, participants experienced a marketplace with e-cigarette liquid prices of $1.63, $3.25, $6.50, and $13.00, while the prices of the other 11 tobacco products remained the same. Units purchased are transformed into mg of nicotine and nonlinear regression is used to estimate the purchasing when e-cigarettes are free/demand intensity, which is reported here. Higher scores indicate more mg of nicotine from e-cigarettes were purchased
Time Frame: 60 minutes post puffing for 4 weeks
Population: All treated and eligible patients
Measure: Mean (95% Confidence Interval); unit: mg of nicotine
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 10 | 10 | 10 | 10
mg of nicotine | 908.3 [425.1 to 2022] | 1142 [539.2 to 2926] | 785.5 [416.1 to 1521] | 985.8 [475.7 to 2416]

9. Other Pre Specified Outcome: Elasticity of Demand or Sensitivity to Price for Each Device Sampled
Description: Demand elasticity , or sensitivity to price, is a behavioral economic measure of of the rate of purchasing decline over increasing cost for e-cigarettes. At each of the four sessions, participants experienced a marketplace with e-cigarette liquid prices of $1.63, $3.25, $6.50, and $13.00, while the prices of the other 11 tobacco products remained the same. Units purchased are transformed into mg of nicotine and nonlinear regression is used to estimate the purchasing when e-cigarettes are free/demand intensity, which is reported here. Higher scores indicate more sensitivity to price, also called inelastic demand.
Time Frame: 60 minutes post puffing for 4 weeks
Population: All treated and eligible patients
Measure: Mean (95% Confidence Interval); unit: mg nicotine per dollar
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 12 | 12 | 12 | 13
mg nicotine per dollar | 0.0005 [.0002 to .0007] | 0.0004 [.0002 to .0006] | 0.0004 [.0002 to .0006] | 0.0005 [.0003 to .0007]

10. Other Pre Specified Outcome: Substitution Levels of Alternative Tobacco Products
Description: Substitution is the slope of the line regressing consumption of the substitute product onto the price of cigarettes (cross-price elasticity). A positive coefficient indicates substitution (use of the substitute increases with increasing cigarette price). A negative value indicates complementarity (use of the substitute declines with increasing cigarette price). A value of 0 indicates no relationship.
Time Frame: 120 minutes post puffing for 4 weeks
Population: All treated and eligible patients
Measure: Mean (95% Confidence Interval); unit: mg nicotine per dollar
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
Number analyzed (Participants) | 10 | 10 | 10 | 10
mg nicotine per dollar
  JUUL Virginia Tobacco | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 7.377 [-0.5177 to 15.27]
  JUUL Classic Tobacco | -0.000000000000 [-87.64 to 87.64] | 8.167 [-69.45 to 85.78] | 2.554 [-81.9 to 87.01] | -4.175 [-95.61 to 87.26]
  JUUL Menthol | 15.54 [-38.02 to 69.11] | 17.31 [-36.31 to 70.93] | 14.75 [-32.1 to 61.61] | 18.28 [-26.91 to 63.47]
  Revel Dark Mint | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Revel Mint | 4.232 [-1.547 to 10.01] | 0.2371 [-2.216 to 2.69] | 4.663 [-0.6079 to 9.935] | 0.2371 [-2.216 to 2.69]
  Marlboro Reds | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Marlboro Menthols | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Camel Snus Mellow | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Camel Snus Frost | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  IQOS Menthol | 4.86 [0.398 to 9.359] | 4.389 [1.230 to 7.548] | 4.432 [-0.622 to 9.485] | 2.43 [-0.9026 to 5.762]
  IQOS Tobacco | 0 [0 to 0] | 0.2552 [-2.385 to 2.895] | 2.382 [-0.1672 to 4.931] | 1.813 [-2637 to 6.262]

ADVERSE EVENTS:
Time Frame: 2 year and 2 months
Arm/Group | A: Unflavored Free-based Nicotine Form | B: Unflavored Salt-based Nicotine Form | C: Tobacco Flavor Free-based Nicotine Form | D: Tobacco Flavor Salt-based Nicotine Form
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT04231539/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT04231539/ICF_001.pdf